CLINICAL TRIAL: NCT06380556
Title: The Effect of Mechanical Vibration and ShotBlocker on Pain Levels During Heel Lance in Healthy Term Neonates: A Randomized Controlled Trial
Brief Title: The Effect of Mechanical Vibration and ShotBlocker on Pain Levels During Heel Lance in Healthy Term Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Aynur Aytekin Ozdemir, Professor, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 25.05.2022/68
Record Dates: First submitted 2024-04-18; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Procedural Pain
Keywords: Procedural pain; Term neonate; Nonpharmacological pain management
MeSH Terms: conditions — Pain, Procedural

STUDY DESIGN:
Intervention Model Description: In the study, participants were assigned to groups by block randomization. Type of delivery (vaginal and cesarean section), gender (male and female) and birth weight (2500-3000 g, 3001-3500 g, 3501 and above) variables were used for block randomization. Blocks were repeated three times in each group and 36 participants were assigned to each. A randomization list with 2 X 2 X 3 X 3 blocks was developed using an online randomization tool. In the study, the group to which the first participant was assigned was determined by a sealed envelope method.
Who Masked: Participant, Outcomes Assessor
Masking Description: Using the block randomization technique, participants were divided into three groups. A web-based randomization list generation tool was used to assign participants to groups. Control and intervention groups were coded as A, B and C using the sealed envelope method. Randomization information was withheld from the researcher involved in data collection until data was collected. The researcher determines which group each baby is in. The researcher found out during the painful procedure. (investigator blinding).
  Within the scope of the research, parents knew which group the baby was in. However, due to the nature of the sample group, the babies were blind.
  To avoid statistical bias, study groups were coded as A, B and C; statistical blinding was performed (statistician blinding).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): The heel lance procedure of the infants in the control group was performed according to the routine heel lance procedure of the clinic.
- ShotBlocker (Experimental): ShotBlocker was applied to the infants in this group before and during the heel lance procedure.
  Interventions: Device: ShotBlocker
- Mechanical vibration (Experimental): Mechanical vibration was applied to the infants in this group before and during the heel lance procedure.
  Interventions: Device: Mechanical vibration

INTERVENTIONS:
Device: ShotBlocker — The protruding surface of the ShotBlocker was placed on the heel lance procedure site. While applying pressure on the skin through the ShotBlocker, the nurse performed heel lancing with the needle through the opening in the center of the ShotBlocker. During the 10-second waiting phase, the ShotBlocker was kept at the procedure site with the same pressure. Then ShotBlocker was removed from the skin and routine capillary blood collection procedure was performed.
  Arms: ShotBlocker
Device: Mechanical vibration — The vibration device was placed on the infant's left extremity in the mid/lateral region just below the knee where the sural nerve passes. The device was secured to the extremity with a gauze bandage. The vibration device was operated for 30 seconds with reference to previous studies. While the vibration continued, the nurse punctured the heel with a needle. Then, the vibration device continued to work in the waiting phase for 10 seconds. The vibration device was removed from the baby's extremity and routine capillary blood collection procedure was performed.
  Arms: Mechanical vibration

SUMMARY:
This study was conducted to determine the effect of mechanical vibration and ShotBlocker methods on pain level, crying time and procedure time during heel prick blood collection in healthy term infants.

DETAILED DESCRIPTION:
Heel prick blood collection, which is one of the painful medical procedures, is one of the diagnostic methods used in newborns and is a more painful procedure compared to other blood collection procedures. Prevention of pain in newborns should be the primary goal of all healthcare personnel working with newborns, both because it is an ethical obligation and because repeated painful exposures have the potential to cause harmful consequences. Nonpharmacologic methods used for the control of acute pain associated with medical procedures are easy to use, have no side effects, are inexpensive and time-saving. Mechanical vibration and ShotBlocker application are among the non-pharmacologic methods frequently used in the management of pain associated with heel prick procedure in term infants.

Previous studies have shown that parent-related methods (kangaroo care, mother/father hug, breastfeeding, etc.) are commonly used for pain management of the newborn during heel prick. In this respect, it is important to determine the effectiveness of mechanical vibration and ShotBlocker methods that can be used independently of the parent, especially in intensive care settings where access to the parent is not always possible.

ELIGIBILITY:
Inclusion Criteria:

* with a postnatal age of 24-72 hours,
* birth weight of 2500 g and above,
* 5th minute APGAR score above 6,
* able to carry out vital activities without support,
* fed within one hour before the procedure,
* calm and not crying before the procedure,
* babies who had heel prick for the first time

Exclusion Criteria:

* with genetic or congenital anomaly,
* with neurological, cardiological and metabolic diseases,
* in need of respiratory support,
* having a history of sedative, analgesic, or narcotic use within 24 h before admission,
* hospitalization and surgical procedure experience in neonatal intensive care unit,
* experience with needle interventions other than vitamin K and Hepatitis B vaccine,
* babies of mothers with a history of substance abuse

Ages: 38 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-07-13 (Actual)

PRIMARY OUTCOMES:
Procedural pain score- Neonatal Infant Pain Scale (NIPS) | 1 min before the heel lance procedure (T-1 min), during the procedure (T+0 sec), 2 min (T+2 min) and 5 min (T+5 min) after the procedure; an average of 6 minutes
  The scale is used to assess procedural pain in neonates. It is a behavioral scale assessing five behavioral indicators (facial expression, cry, arms, legs, and state of alertness) and one physiological indicator (breathing patterns). Five items (facial expression, breathing pattern, arms, legs, and state of alertness) are scored as 0 (Good) or 1 (Bad), while one item (crying) is scored as 0 (Good), 1, or 2 (Bad). The total scale score ranges from 0 to 7, with higher scores indicating more pain.

SECONDARY OUTCOMES:
Crying time | Through painful procedure completion, an average of 5 minutes
  Crying time is the crying time between the moment of heel puncture and 5 minutes after the procedure.
Procedure time | Through painful procedure completion, an average of 2 minutes
  The duration of the procedure is the time between the moment of heel lance and the closure of the heel with gauze after the collection of capillary blood.

CONTACTS AND LOCATIONS:
Overall Officials: Aynur Aytekin Özdemir, PhD, Study Director — Istanbul Medeniyet University
Locations (1):
- Istanbul Medeniyet University, Istanbul, Kadıköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be shared upon request from the principal investigator, subject to the appropriateness of the request, while ensuring adherence to the rules of confidentiality regarding individual data.
Supporting Information: Study Protocol
Time Frame: September through December of 2025
Access Criteria: Individual participant data may be shared upon request from the principal investigator, subject to the appropriateness of the request, while ensuring adherence to the rules of confidentiality regarding individual data.

REFERENCES:
- [Background] Avan Antepli N, Bilsin Kocamaz E, Gungormus Z. The Effect of Vibration on Pain During Heel Lance Procedures in Newborns: A Randomized Controlled Trial. Adv Neonatal Care. 2022 Apr 1;22(2):E43-E47. doi: 10.1097/ANC.0000000000000918. PMID 34334677
- [Background] McGinnis K, Murray E, Cherven B, McCracken C, Travers C. Effect of Vibration on Pain Response to Heel Lance: A Pilot Randomized Control Trial. Adv Neonatal Care. 2016 Dec;16(6):439-448. doi: 10.1097/ANC.0000000000000315. PMID 27533335
- [Background] Baba LR, McGrath JM, Liu J. The efficacy of mechanical vibration analgesia for relief of heel stick pain in neonates: a novel approach. J Perinat Neonatal Nurs. 2010 Jul-Sep;24(3):274-83. doi: 10.1097/JPN.0b013e3181ea7350. PMID 20697246
- [Background] Caglar S, Buyukyilmaz F, Cosansu G, Caglayan S. Effectiveness of ShotBlocker for Immunization Pain in Full-Term Neonates: A Randomized Controlled Trial. J Perinat Neonatal Nurs. 2017 Apr/Jun;31(2):166-171. doi: 10.1097/JPN.0000000000000256. PMID 28437308
- [Derived] Catal RA, Ozdemir AA, Karatekin G. Effect of mechanical vibration and ShotBlocker(R) on pain levels during heel lance in healthy term neonates: A randomized controlled trial. J Pediatr Nurs. 2024 Nov-Dec;79:e51-e59. doi: 10.1016/j.pedn.2024.09.019. Epub 2024 Oct 11. PMID 39394025